CLINICAL TRIAL: NCT01483911
Title: Phase I, Single-centre, Randomised, Placebo-controlled, Double-blinded Study, With Single Ascending Dose and Multiple Dose at Maximum Tolerated Dose, Evaluating the Safety, Tolerability and Pharmacokinetics of ALX-0171, Administered by Pulmonary Inhalation, in Healthy Male Volunteers
Brief Title: ALX-0171 Phase I Study, Evaluating Single Ascending Dose and Multiple Dose in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ablynx, a Sanofi company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALX-0171-1.1/11
Record Dates: First submitted 2011-11-30; First posted 2011-12-02 (Estimated); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: RSV Infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — gontivimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ALX-0171 (Experimental)
  Interventions: Biological: ALX-0171
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: ALX-0171 — Single or multiple ascending doses (2.1-210 mg), administered via pulmonary inhalation. Multiple dosing will consist of twice daily dosing on 5 consecutive days.
  Arms: ALX-0171
Biological: Placebo — Single or multiple doses, administered via pulmonary inhalation. Multiple dosing will consist of twice daily dosing on 5 consecutive days.
  Arms: Placebo

SUMMARY:
ALX-0171 is a Nanobody directed against the human respiratory syncytial virus (RSV). The purpose of this first-in-man study is to determine the safety, tolerability and pharmacokinetics (PK) of ALX-0171 after single and multiple pulmonary administrations in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking healthy male volunteers, aged 18-55 years
* Good health condition, as determined by medical history, physical examination and clinical laboratory testing
* Forced expiratory volume in 1 second (FEV1) ≥ 90% of predicted value
* Diffusing capacity of the lung for CO (DLCO) ≥ 85% of predicted value
* Normal chest X-Ray (anteroposterior and lateral view)
* Minimum weight of 70.0 kg, minimum height of 1m70, body mass index between 18.0 and 30.0 kg/m²

Exclusion Criteria:

* Current smokers, or ex-smokers abstinent from tobacco for less than one year
* History or presence of atopy or pulmonary non-specific hyperreactivity
* Positive bronchial challenge test
* Symptomatic viral infection, or suspicion thereof (including rhinitis) in last 14 days prior to dosing
* Signs of active pulmonary infection or other inflammatory conditions, even in the absence of febrile episodes, in the last 14 days prior to dosing

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
number of treatment-emergent adverse events | until 1 month after last study drug administration

SECONDARY OUTCOMES:
plasma concentration of ALX-0171 | from predose until 5 days after study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Josefin-Beate Holz, MD, Study Director — Ablynx, a Sanofi company
Locations (1):
- Groningen, Netherlands